CLINICAL TRIAL: NCT03423563
Title: Comparison of Endotracheal Intubation Using Flexible Fiberoptic Bronchoscopy Versus Flexible Intubation Video Endoscope (FIVE) in Obese Patients Undergoing Elective Surgeries Under General Anesthesia: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Mohamed, Ahmed A., M.D. (Individual); Mai Wedad Ahmed (Unknown); Norhan Abdelaleem Ali (Unknown); Magdy Abdelmohsen Elsayed (Unknown); Atef Kamel Salama (Unknown)
Responsible Party: Principal Investigator, Ahmed Abdalla, Assistant Professor of Anesthesia&I.C.U and Pain Clinic, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: N-68-2016/Ms
Record Dates: First submitted 2017-12-26; First posted 2018-02-06 (Actual); Last update posted 2018-03-16 (Actual); Status verified 2018-03

CONDITIONS: Flexible Fiberoptic Bronchoscopy Versus Flexible Intubation Video Endoscope FIVE in Obese Patients

STUDY DESIGN:
Intervention Model Description: In this prospective randomized controlled study 60 patients with ASA physical status Ӏ-ӀӀ, aging 20-50 years will be randomly allocated into two groups, 30 patients in each group
Masking Description: In this prospective randomized controlled study 60 patients with ASA physical status Ӏ-ӀӀ, aging 20-50 years will be randomly allocated into two groups, 30 patients in each group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Flexible fiberoptic bronchoscopy (Experimental): Fiberoptic intubation has been considered for a long time the gold standard technique for intubation when there is anticipated or known difficult airway or as a rescue device in can't intubate but can ventilate scenarios
  Interventions: Device: Flexible fiberoptic bronchoscopy
- Fexible intubation video endoscopy (Experimental): Video-assisted techniques allow to indirectly visualize the laryngeal structures with fiber optical or camera chip technique and to show the video picture on an external or built-in monitor
  Interventions: Device: Fexible intubation video endoscopy

INTERVENTIONS:
Device: Flexible fiberoptic bronchoscopy — Flexible fiberoptic bronchoscopy versus flexible intubation video endoscope regarding intubation time in obese patients
  Arms: Flexible fiberoptic bronchoscopy
Device: Fexible intubation video endoscopy — Fexible intubation video endoscopy
  Arms: Fexible intubation video endoscopy

SUMMARY:
Tracheal intubation is one of the most common medical procedures performed in hospitals. On one hand, it is highly successful and easy to perform using a rigid laryngoscope. On the other hand, hypoxic brain damage and death may result rapidly if it is unsuccessful. This disastrous outcome happens when the airway cannot be secured by intubation and face mask ventilation becomes difficult.

Careful preoperative evaluation to identify patients in whom tracheal intubation and mask ventilation may prove to be difficult can save lives.

Over the past 40 years, different techniques of tracheal intubation have been introduced, the most effective under different conditions being fiberoptic intubation.

The flexible intubation video endoscope is a relatively new device which delivers clear, pixel-free images without a Moiré pattern. The flexible intubation video endoscope can be directly connected to the C-MAC® monitor. Due to the Distal Chip technology the user enjoys a full-format direct video imaging with improved image quality with a resolution higher than fiberoptic bronchoscopy which has another disadvantage of being Fragile where Fibres can be broken or have transmission loss when wrapped around curves of only a few centimeters radius.

After ethics approval and informed consent from patients, 60 obese patients aging from 20-60 years will randomly allocated and divided into two groups each is (Thirty) patients in each group, using flexible intubation video endoscope(FIVE) in (group1) and fiberoptic bronchoscopy in (group 2).

The study will compare the techniques for time of intubation, hemodynamic (SBP, DBP and HR) changes, success rate, number of attempts and complications in both groups.

investigators expect from this study that flexible intubation video endoscope(FIVE) has become a good alternative and associated with better visualization of laryngeal structures in shorter time as compared to traditional flexible fiberoptic bronchoscopy.

DETAILED DESCRIPTION:
Airway management is considered a cardinal aspect of anesthetic practice and of emergency and intensive care medicine. Endotracheal intubation is a simple, safe, rapid and nonsurgical method that achieves all the objectives of airway management which include maintaining a patent airway, lung protection from aspiration and allows leak free ventilation during mechanical ventilation. Even though endotracheal intubation isn't a complication free procedure, some of them life-threatening. It is important to anesthesiologists to be alert to these complications and to have an effective plan to avoid and manage these complications when they occur .

If a clear airway can't be guaranteed, it can be fatal. In 1990, an analysis of anesthesia-related closed claims in the USA declared that respiratory system adverse outcomes were the lone largest class of injury and that the percentage of death or catastrophic brain insult associated with it was much higher than that associated with cardiovascular problems.Since then, it became a priority to decrease the serious adverse outcomes associated with airway management; major protocols for difficult airway management have been defined, developing new reliable airway devices, and adequate monitoring of ventilation by pulse oximetry and capnography have become a standard. Thanks to these efforts, the incidence of these serious adverse outcomes is likely to be reduced, and airway management can now be considered as a safe procedure.

Endotracheal intubation is still the "gold standard" in airway management . If with using traditional techniques or video-assisted techniques which can be used when there is intubation failure or anticipated difficult airway. Video-assisted techniques may help to increase intubation success.

Video-assisted techniques allow to indirectly visualize the laryngeal structures with fiber optical or camera chip technique and to show the video picture on an external or built-in monitor.

Fiberoptic intubation has been considered for a long time the gold standard technique for intubation when there is anticipated or known difficult airway or as a rescue device in can't intubate but can ventilate scenarios . Fibreoptic intubation can be a hard skill to teach, gain and keep.In this context, closed claims analysis has declared severe complications such as catastrophic brain insult and death occurred with anticipated difficult airway management and awake intubation. Therefore, it is considerable to develop simple, dependable, safe, and effective intubation devices.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 and 50 years.
* Scheduled for elective surgery requiring endotracheal intubation.
* Patient with ASA physical status I-II.

Exclusion Criteria:

* • Unable to give consent

  * Patient with ASA physical status more than II.
  * Age < 20years old and >50years
  * Pregnant patient.
  * Known, difficult airway
  * Loose teeth
  * Require a rapid sequence induction,
  * If special endotracheal tube (ETT) is needed for the case.
  * Emergency surgeries

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-01-04 (Actual); Primary Completion 2018-02-05 (Actual); Study Completion 2018-02-11 (Actual)

PRIMARY OUTCOMES:
Successful intubation | Intraoperative
  Time in Minutes of successful intubation.

SECONDARY OUTCOMES:
Rate of first successful intubation | Intraoperative
  Rate of first time success intubation
Second trial for successful intubation | Intraoperative
  Intubation success in second trial

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Abdalla Mohamed, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
Via scholar Gate